CLINICAL TRIAL: NCT06365307
Title: Non-Randomized Controlled Comparative Study of Gene-Activated Osteoplastic Material "Histograft" in Patients With Degenerative Diseases of the Lumbar and Cervical Spine
Brief Title: Comparative Study of Gene-Activated Bone Substitute "Histograft" for Lumbar and Cervical Spinal Fusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Histograft Co., Ltd. (Industry)
Collaborators: Petrovsky National Research Center of Surgery (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Histograft-SF-2023
Record Dates: First submitted 2024-04-08; First posted 2024-04-15 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-04

CONDITIONS: Cervical Disc Disorder With Radiculopathy; Spinal Stenosis; Lumbar and Other Intervertebral Disc Disorders With Radiculopathy; Biomechanical Lesion, Unspecified
Keywords: Spinal fusion; Bone graft
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: During the preliminary screening and indication for surgical treatment, patients are divided into 2 groups depending on the location of the pathological process: 1 - cervical spine, 2 - lumbar spine. During independent sequential randomization in a 1:1 ratio, patients in each of these groups are divided into clinical (A) and control (B) groups.
  Distribution of treatment methods by groups:
  1A - use of "Histograft" for spinal fusion of the cervical spine, 50 patients
  1. B - use of synthetic osteoplastic material based on β-TCP for spinal fusion of the cervical spine, 50 patients
  2. A - use of "Histograft" for spinal fusion of the lumbar spine, 100 patients
  2B - use of bone autograft for spinal fusion of the lumbar spine, 100 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical group (Experimental): Group of patients, who is treated with usage of Histograft bone substitute (gene-activated matrix based on octacalcium phosphate and plasmid DNA encoding VEGFA gene) in spinal fusion of cervical or lumbal spine
  Interventions: Combination Product: Osteoplastic material based on octacalcium phosphate and biologically active nucleic acids for bone tissue regeneration Nucleostim-VEGF ("Histograft")
- Control group (Active Comparator): Group of patients, who get standard treatment with usage of synthetic osteoplastic material based on β-TCP for spinal fusion of the cervical spine or use of bone autograft for spinal fusion of the lumbar spine
  Interventions: Other: Synthetic osteoplastic material based on β-TCP or bone autograft

INTERVENTIONS:
Combination Product: Osteoplastic material based on octacalcium phosphate and biologically active nucleic acids for bone tissue regeneration Nucleostim-VEGF ("Histograft") — Due to the localization of the pathological process, all patients are divided into two groups: 1 - cervical spine, 2 - lumbar spine. Within these groups, patients are treated with either gene-activated osteoplastic material Histograft or synthetic osteoplastic material based on β-TCP (β-tricalcium phosphate) for spinal fusion of the cervical spine, or with bone autograft for spinal fusion of the lumbar spine.
  Arms: Clinical group
Other: Synthetic osteoplastic material based on β-TCP or bone autograft — Due to the localization of the pathological process, all patients are divided into two groups: 1 - cervical spine, 2 - lumbar spine. Within these groups, patients are treated with either gene-activated osteoplastic material Histograft or synthetic osteoplastic material based on β-TCP (β-tricalcium phosphate) for spinal fusion of the cervical spine, or with bone autograft for spinal fusion of the lumbar spine.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of the combination product "Histograft", a bone substitute based on octacalcium phosphate (OCP) and plasmid DNA encoding VEGFA gene, in spinal fusion prosedure in comparison with bone autografts and synthetic material based on β-TCP

DETAILED DESCRIPTION:
An open-label non-randomized controlled clinical trial will be conducted with two groups of patients. Following enrollment based on specific indication criteria, all patients will undergo surgical treatment (spinal fusion) using either bone substitute "Histograft" (for spinal fusion of cervical and lumbar spine) or bone autograft (for spinal fusion of lumbar spine), or synthetic material based on β-TCP (for spinal fusion of cervical spine). The primary outcomes will involve the bone fusion rate evaluated with computer tomography (CT) at 6 and 12 months. For the safety assessment, the frequency of serious adverse events (SAEs) and adverse events (AEs) will be monitored throughout the entire clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* signing the informed consent
* indications for spinal fusion: degenerative-dystrophic diseases of the cervical and lumbar spine.

Exclusion Criteria:

* refusal to sign IP
* age less than 18 years
* history of spinal surgery in the area of planned spinal fusion
* decompensated forms of chronic diseases
* oncological diseases with identified metastases or risk of metastasis
* patient's refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Spinal fusion | 6 and 12 months after intervention
  Vertebral fusion: formation of a "bone block" according to CT data (regenerated bone density between the vertebrae without areas of fibrosis and signs of resorption around metal structures)
Adverse events and Severe Adverse Events | Within 1 year after intervention
  Frequency of Adverse and Severe Adverse Events after treatment

SECONDARY OUTCOMES:
SF- 36 score (The Short Form-36) | 6 and 12 months after treatment
  Assessment of life quality. A score value is ranging from 0 to 100. Higher scores indicate better health status
Unexpected Adverse Drug Reaction | Within 1 year after intervention
  Identification of Unexpected Adverse Drug Reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Clinical Center No. 2 of Federal State Budgetary Research Institution "Russian research center of surgery named after academician B.V.Petrovsky", Moscow, Moscow Oblast, Russia

IPD SHARING:
Plan to Share IPD: No